CLINICAL TRIAL: NCT01244516
Title: Multi-Center 2-Week Clinical Evaluation of Three Silicone Hydrogel Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CR-201007
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-04

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- galyfilcon A (Other): Subjects that were randomized to receive the galyfilcon A lens with a base curve of 8.30 throughout the entire course of the study.
  Interventions: Device: galyfilcon A, BC 8.30
- lotrafilcon B (Other): Subjects that were randomized to wear lotrafilcon B lens throughout the course of the study.
  Interventions: Device: lotrafilcon B, BC 8.60
- comfilcon A (Other): Subjects that were randomized to wear comfilcon A lens throughout the course of the study.
  Interventions: Device: comfilcon A, BC 8.60

INTERVENTIONS:
Device: galyfilcon A, BC 8.30 — galyfilcon A, BC 8.30 soft contact lens
  Arms: galyfilcon A
Device: lotrafilcon B, BC 8.60 — lotrafilcon B, BC 8.60 soft contact lens
  Arms: lotrafilcon B
Device: comfilcon A, BC 8.60 — comfilcon A, BC 8.60 soft contact lens
  Arms: comfilcon A

SUMMARY:
The purpose of this study is to compare the clinical performance of three silicone hydrogel contact lenses over a 2 week period.

ELIGIBILITY:
Inclusion Criteria:

* Be no less than 18 and no more than 39 years of age.
* Sign Written Informed Consent and investigator to record this on Case Report Form.
* Be willing and able to adhere to the instructions set out in the protocol.
* Be an existing successful daily wear soft contact lens wearer. For the purposes of this study this means wearing lenses for at least 6 hours per day, 5 days per week for the last month.
* No extended wear in the last 3 months.
* Subjective refraction must result in a vertex corrected spherical contact lens prescription between -1.00 and -6.00 diopters.
* Have refractive astigmatism less than or equal to 1.00 diopters (D) in both eyes.
* Achieve visual acuity of 6/9 (20/30) or better in each eye.
* Require a visual correction in both eyes (no monovision allowed).
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having: no amblyopia, no evidence of lid abnormality or infection (including blepharitis/meibomitis), no conjunctival abnormality or infection, no clinically significant slit lamp findings (i.e. stromal edema, vascularization, infiltrates or abnormal opacities), no other active ocular disease.

Exclusion Criteria:

* Requires concurrent ocular medication.
* Clinically significant corneal stromal haze, corneal vascularization, tarsal abnormalities, bulbar hyperemia, limbal hyperemia, or any other abnormality of the cornea that would contraindicate contact lens wear.
* Clinically significant corneal staining
* Requires presbyopic correction (i.e. Not using any presbyopic correction and measured add power of less than +1.00 diopters).
* Has had refractive surgery.
* Has had eye injury/surgery within 8 weeks immediately prior to enrollment for this study.
* Abnormal lacrimal secretions.
* Pre-existing ocular irritation that would preclude contact lens fitting.
* Keratoconus or other corneal irregularity.
* Hard, hybrid or Rigid Gas Permeable lens wear in the previous 8 weeks.
* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Diabetic.
* Infectious disease (e.g., hepatitis, tuberculosis) or an immunosuppressive disease [e.g., Human immunodeficiency virus (HIV)].
* History of chronic eye disease (e.g. glaucoma or Age Related Macular Degeneration).
* Pregnancy, lactating or planning a pregnancy at the time of enrollment.
* Participation in any concurrent clinical trial or in last 30 days

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 540 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (34):
- United States (34):
  - Brea, California
  - Campbell, California
  - Cupertino, California
  - Mission Viejo, California
  - Colorado Springs, Colorado
  - Bridgeport, Connecticut
  - Aventura, Florida
  - Jacksonville, Florida
  - Tallahassee, Florida
  - Tampa, Florida
  - Winter Park, Florida
  - Roswell, Georgia
  - Bloomington, Illinois
  - Mishawaka, Indiana
  - Pittsburg, Kansas
  - Boston, Massachusetts
  - Independence, Missouri
  - Raytown, Missouri
  - Closter, New Jersey
  - New York, New York
  - Raleigh, North Carolina
  - North Olmsted, Ohio
  - Powell, Ohio
  - Kittanning, Pennsylvania
  - Warwick, Rhode Island
  - Chamberlain, South Dakota
  - Bartlett, Tennessee
  - Brentwood, Tennessee
  - Memphis, Tennessee
  - Tyler, Texas
  - Salt Lake City, Utah
  - Burlington, Vermont
  - Salem, Virginia
  - Virginia Beach, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were thirty-five sites recruited in the US. There were 540 subjects recruited with 520 enrolled and randomized. The study was a 2-week, randomized, single-masked (subjects), parallel arm, bilateral dispensing study. The subject group was expected to be representative of a cross-section of the population within the US contact lens market.
Pre-assignment Details: There were 20 subjects who did not meet the inclusion or did meet the exclusion criteria. There were 10 screen failures and 10 who wore spectacles to baseline visit invoking the exclusion criteria.
Period: Period 1 (Baseline to 1-week Visit)
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A
Started | 170 | 177 | 173
Completed | 166 | 171 | 170
Not Completed | 4 | 6 | 3
Not completed — Protocol Violation | 4 | 5 | 2
Not completed — Poor Vision | 0 | 1 | 0
Not completed — Poor comfort | 0 | 0 | 1
Period: Period 2 (1-week to 2-week Visit)
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A
Started | 166 | 171 | 170
Completed | 163 | 170 | 168
Not Completed | 3 | 1 | 2
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 1
Not completed — Lost to Follow-up | 0 | 1 | 0
Not completed — Poor Comfort | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Population consists of those subjects who were enrolled and randomly assigned to a treatment arm AND who completed the study per protocol.
Groups:
- Total: Total of all reporting groups
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A | Total
Number analyzed (Participants) | 163 | 170 | 168 | 501
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.8 (5.9) | 28.3 (5.6) | 27.4 (5.7) | 28.2 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 118 | 115 | 341
  Male | 55 | 52 | 53 | 160
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 163 | 170 | 168 | 501

OUTCOME MEASURES:

1. Primary Outcome: Overall Subjective Comfort
Description: Contact Lens User Experience (CLUE)TM questionnaire: A validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response.
Time Frame: after 2 weeks of contact lens wear
Population: Analysis is on those subjects who completed the study (n=501).
Measure: Least Squares Mean (Standard Error); unit: CLUE score
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 163 | 170 | 168
CLUE score | 51.7 (2.1) | 51.3 (2.0) | 51.3 (2.0)
Statistical Analysis 1: Comparison: Galyfilcon A vs Lotrafilcon B; This comparison is between galyfilcon and lotrafilcon B. Ho: galyfilcon A -lotrafilcon B <= -5. Ha: galyfilcon A - lotrafilcon B > -5; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is set at -5; Mixed Models Analysis; Alpha is adjusted to 1.3% based on a Sidak multiplicity correction; Mean Difference (Final Values) = 0.39, 97.4% CI 2-sided [-5.91 to 6.70], Standard Error of Mean 2.83 — The direction of comparison is AAHP - AOA
Statistical Analysis 2: Comparison: Galyfilcon A vs Comfilcon A; This comparison is between galyfilcon A and comfilcon A. Ho: gayfilcon A- comfilcon A <= -5. Ha: galyfilcon A- comfilcon A> -5; Test type: Non-Inferiority or Equivalence — The non-inferiority margin is set at -5; Mixed Models Analysis; Alpha is adjusted to 1.3% based on a Sidak multiplicity correction; Mean Difference (Final Values) = 0.42, 97.4% CI 2-sided [-5.96 to 6.79], Standard Error of Mean 2.79 — The direction of comparison is AAHP - BIO

2. Primary Outcome: Corneal Staining
Description: Investigator evaluated corneal staining. Percent of eyes with corneal staining presence or absence is evaluated.
Time Frame: after 2 weeks of contact lens wear
Population: Analysis is on those subjects who completed the study (n=501).
Measure: Number; unit: percentage of eyes
Units Other Than Participants: Eyes
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A
Number analyzed (Participants) | 163 | 170 | 168
Number analyzed (Eyes) | 326 | 340 | 336
percentage of eyes
  No corneal staining | 78.5 | 67.1 | 66.1
  With corneal staining | 21.5 | 32.9 | 33.9
Statistical Analysis 1: Comparison: Galyfilcon A vs Lotrafilcon B; The comparison is between galyfilcon A (AAHP) and lotrafilcon B (AOA) for comparing proportions of those with corneal staining and those without. Ho: OR = 1 for (AAHP/AOA). Ha: OR > 1 for (AAHP/AOA); Test type: Non-Inferiority or Equivalence — The non-inferiority margin is set at > 0.75. Superiority is concluded is the 97.4% CL > 1; Regression, Logistic; Alpha is adjusted to 1.3% based on a Sidak multiplicity correction; Odds Ratio (OR) = 1.66, 97.4% CI 2-sided [1.14 to 2.44] — The direction of comparison is AAHP/AOA
Statistical Analysis 2: Comparison: Galyfilcon A vs Comfilcon A; The comparison is between galyfilcon A (AAHP) and comfilcon A (BIO) for comparing proportions of those with corneal staining and those without. Ho: OR = 1 for (AAHP/BIO). Ha: OR > 1 for (AAHP/BIO); Test type: Non-Inferiority or Equivalence — The non-inferiority margin is set at > 0.75. Superiority is concluded is the 97.4% CL > 1; Regression, Logistic; Alpha is adjusted to 1.3% based on a Sidak multiplicity correction; Odds Ratio (OR) = 1.66, 97.4% CI 2-sided [1.14 to 2.44]

3. Secondary Outcome: Overall Subjective Lens Handling
Description: Contact Lens User Experience (CLUE)TM questionnaire: A validated patient-reported outcomes questionnaire to assess patient-experience attributes of soft, disposable contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Scores follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0 to 120. Only galyficlon A and comfilcon A were evaluated.
Time Frame: after 2 weeks of contact lens wear
Population: Analysis is on those subjects who completed the study (n=331) and where assigned to these two arms. Analysis is restricted to these two arms for this outcome as specified per protocol.
Measure: Least Squares Mean (Standard Error); unit: CLUE score
Arm/Group | Galyfilcon A | Comfilcon A
Number analyzed (Participants) | 163 | 168
CLUE score | 64.3 (1.6) | 59.8 (1.6)

ADVERSE EVENTS:
Arm/Group | Galyfilcon A | Lotrafilcon B | Comfilcon A
Serious Adverse Events (participants affected / at risk) | 0/170 | 0/177 | 0/173
Other Adverse Events (participants affected / at risk) | 0/170 | 0/177 | 0/173

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication required agreement and written authorization from the Sponsor.